CLINICAL TRIAL: NCT05138003
Title: Detection of Myocardial Inflammation in Cyclists After Strenuous Exercise: a Pilot Study Part 2
Brief Title: COUREUR Study Myocardial Inflammation in Cyclist Part 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Collaborators: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021/051
Record Dates: First submitted 2021-06-18; First posted 2021-11-30 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Myocardial Inflammation
MeSH Terms: conditions — Myocarditis | interventions — Echocardiography; Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recreational cyclists performing the 'étape du tour (EDT) de France 2021 (Other)
  Interventions: Diagnostic Test: cardiac MRI; Diagnostic Test: Echocardiography; Diagnostic Test: RootiRx for the ECG monitoring during the cycling ride; Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: cardiac MRI — T1 and T2 relaxation times will be evaluated on basal and mid-cavity SA maps; a single ROI measurement in the septum will be manually drawn sufficiently far from tissue interfaces to avoid the impact of susceptibility artifacts from adjacent tissues. The differences in T1 and T2 relaxation times between rest and post-exercise will be analyzed.
  Cardiac ventricular volumes, function and LV mass will also be quantified.
Diagnostic Test: Echocardiography — Measurements of mass, volumes and function will be obtained of both the left and right ventricles enabling comparisons with cardiac MRI and traditional echo measures.
Diagnostic Test: RootiRx for the ECG monitoring during the cycling ride — The final report will include the amount of recorded beats, the average heart rate, the maximum and minimum heart rate, the amount of cardiac pauses defined as an interruption in the ventricular rate > 2 seconds. Reported atrial events include atrial ectopic beats and supraventricular tachycardia and ventricular events include ventricular ectopic beats, doublets, triplets, bigeminy, trigeminy and ventricular tachycardia.
Diagnostic Test: Blood sample — Blood sample will be performed 3 to 6 hours after the stage to analyze high-sensitivity cardiac Troponin T (high-sensitivity) levels, Creatine Phosphokinase (CPK) to eliminate the hypothesis of Troponin elevation induced by rhabdomyolysis and C-reactive Protein to corroborate the inflammatory aspect if there is any.

SUMMARY:
The study will evaluate myocardial inflammation in cyclists after high intense and sustained exercise. Our hypothesis is that strenuous exercise in recreational cyclists may be associated with myocardial inflammation. Myocardial fibrosis in asymptomatic athletes is associated with life-threatening arrhythmic events and sudden death. Although myocarditis seems to be the most likely underlying cause, it remains unclear if strenuous and sustained physical exercise can cause myocardial inflammation with development of myocyte necrosis and possibly myocardial fibrosis in athletes.

Nineteen recreational cyclists performing "L'ETAPE DU TOUR (EDT) de France" a cycling ride (175 km, 3600 m of positive altitude difference) on July 4 2021 will be included in this study. Each participant will complete a detailed questionnaire detailing their training history. All participants will have exercise testing approximately 1 week before the EDT stage to set aerobic and anaerobic gas exchange thresholds, as well as VO2max.

In part 2 of the study cardiac MRI will be performed at rest before the EDT cycling ride completion. An ECG registration using a RootiRx will be realized during and up to 6 hours after the cycling ride. An echocardiography and cardiac MRI will be repeated in each cyclist between 3 and 6 hours after EDT cycling ride completion. A blood sample will be obtained at that time after the ride. This time point is chosen based on the highest troponin release that 3 to 6 hours post-exercise would allow a sufficient amount of time for inflammation to develop and be detectable, corresponding with the time when cardiac Troponin T is typically detectable and representing the liberation of enzymes from damaged myocytes.

Finally, a third cardiac MRI will be repeated 24 hours after start of the cycling ride to verify the evolution of possible inflammation over this time period.

ELIGIBILITY:
Inclusion Criteria:

* Recreational cyclists performing the 'étape du tour (EDT) de France 2021 ride

Exclusion Criteria:

* presence of pre-existing cardiovascular or pulmonary diseases, hypertension, diabetes, peripheral vascular diseases, any inflammatory or auto-immune diseases, active SARS-CoV-2 infection and the intake of anti-inflammatory drugs.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Myocardial inflammation will be evaluated by T1/T2 mapping cardiac MRI in cyclists after a strenuous exercise | 12 months after study
  T1 and T2 relaxation time will be measured on cardiac MRI in cyclists before and 3 to 6 hours after a high intense and sustained exercise to assess exercise-induced myocardial inflammation

CONTACTS AND LOCATIONS:
Locations (2):
- Jessa Hospital, Hasselt, Belgium
- Centre Hospitalier Universitaire de Nice, Nice, France

REFERENCES:
- [Derived] Ghekiere O, Herbots L, Peters B, Berg BV, Dresselaers T, Franssen W, Padovani B, Ducreux D, Ferrari E, Nchimi A, Demanez S, De Bosscher R, Willems R, Heidbuchel H, La Gerche A, Claessen G, Bogaert J, Eijnde BO. Exercise-induced myocardial T1 increase and right ventricular dysfunction in recreational cyclists: a CMR study. Eur J Appl Physiol. 2023 Oct;123(10):2107-2117. doi: 10.1007/s00421-023-05259-4. Epub 2023 Jul 22. PMID 37480391